CLINICAL TRIAL: NCT05985252
Title: Virtual Ileostomy Versus Conventional Loop Ileostomy in Patients Undergoing Low Anterior Resection for Rectal Cancer: A Randomized Controlled Study
Brief Title: Virtual Ileostomy Versus Conventional Loop Ileostomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, fan li, Professor, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-RCT
Record Dates: First submitted 2023-07-14; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Rectal Neoplasms
Keywords: Virtual ileostomy; Diverting ileostomy; Rectal Neoplasms; Rectosigmoid junction
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual ileostomy (Experimental): Laparoscopic or robotic surgery with virtual ileostomy
  Interventions: Procedure: Virtual ileostomy
- Diverting ileostomy (Active Comparator): Laparoscopic or robotic surgery with diverting ileostomy
  Interventions: Procedure: Diverting ileostomy

INTERVENTIONS:
Procedure: Virtual ileostomy — Laparoscopic or robotic surgery with virtual ileostomy
  Arms: Virtual ileostomy
Procedure: Diverting ileostomy — Laparoscopic or robotic surgery with diverting ileostomy
  Arms: Diverting ileostomy

SUMMARY:
This study aimed at comparing the Comprehensive Complication Index (CCI), readmission rates, postoperative hospitalization days, duration of bearing the stoma (months), hospitalization costs, the number of hospitalizations with ghost ileostomy versus conventional loop ileostomy after low anterior resection for rectal cancer.

DETAILED DESCRIPTION:
Diverting ileostomy (DI) is a common procedure performed in patients undergoing low anterior resection for rectal cancer to protect the anastomosis and reduce the risk of complications. Although DI remains one of the most common methods used in clinical practice to prevent anastomotic leakage, there is still considerable debate in clinical practice about whether to perform a routine ileostomy. Despite temporary ileostomy fecal diversion can reduce the development of abdominal abscesses, wound inflammation, peritonitis, and sepsis after the occurrence of AL, however, it not only failed to reduce the incidence of AL but significantly increased the risk of non-elective readmissions and reinterventions as well as higher total costs. Meanwhile, stoma significantly increase the risk of stoma-related complication such as small bowel obstruction, postoperative ileus, dehydration from high-output stoma culminating in acute kidney injury, electrolyte imbalance, stoma stenosis/ necrosis, parastomal hernia, peristomal abscess, and fistula, etc.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed low to intermediate level rectal cancer, with the lower margin of anastomosis <10cm from the anus.
* age ≥18 years and ≤80 years.
* the surgical procedure is anterior rectal resection (LAR).
* intraoperative virtual or conventional ileostomy was performed.

Exclusion Criteria:

* BMI >30 kg/m².
* ASA score >3.
* Patients with coexisting complete intestinal obstruction.
* History of long-term use of immunosuppressive drugs or glucocorticoids.
* Combined severe cardiac disease: with congestive heart failure or NYHA cardiac function ≥ grade 2. Patients with a history of myocardial infarction or coronary artery surgery within 6 months prior to the procedure.
* chronic renal failure (requiring dialysis or glomerular filtration rate <30 mL/min).

Intraoperative combined multi-organ resection.

* Combined cirrhosis of the liver.
* Intraoperative findings of incomplete anastomosis and positive insufflation test.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Calculation postoperative of the Comprehensive Complication Index (CCI) for each patient | An average of 1 year from the date of low anterior resection for rectal cancer until the date of when the patient's condition is stabilized without complications
  The Comprehensive Complication Index (CCI)summarises all postoperative complications based on the established Clavien-Dindo classification (ranging from mild complications not leading to a deviation from the normal clinical course (grade I) up to postoperative death (grade V)) at an individual patient level according to their grade of severity.

SECONDARY OUTCOMES:
Postoperative hospitalization days | Through study completion, an average of 1 year
  Patients in the virtual stoma group who did not have a second surgery due to complications recorded days of postoperative hospitalization after low anterior resection for rectal cancer, if the virtual stoma group required bedside or secondary surgery for diverting ileostomy due to complications and all patients in the diverting ileostomy group required reoperation for stoma reversal, record days of postoperative hospitalization due to complications and/or reoperation since the data of low anterior resection for rectal cancer.
Readmission rates | Through study completion, an average of 1 year
  Patients in the virtual stoma group who did not have a second surgery due to complications recorded the number of hospitalization after low anterior resection for rectal cancer. If the virtual stoma group required bedside or secondary surgery for diverting ileostomy due to complications and all patients in the diverting ileostomy group required reoperation for stoma reversal, record the number of hospitalization due to complications and/or reoperation since the data of low anterior resection for rectal cancer.
The number of hospitalizations | Through study completion, an average of 1 year
  Patients in the virtual stoma group who did not have a second surgery due to complications recorded the number of hospitalization after low anterior resection for rectal cancer. If the virtual stoma group required bedside or secondary surgery for diverting ileostomy due to complications and all patients in the diverting ileostomy group required reoperation for stoma reversal, record the number of hospitalization due to complications and/or reoperation since the data of low anterior resection for rectal cancer.
Duration of bearing the stoma (months) | Through study completion, an average of 1 year
  If the virtual stoma group required bedside or secondary surgery for diverting ileostomy due to complications and all patients in the diverting ileostomy group required reoperation for stoma reversal, record the duration of bearing the stoma since the data of surgery of diverting ileostomy.
First hospitalization costs | During hospitalization,approximately 7 days
  Patient hospitalization costs for radical resection of rectal cancer.
Total hospitalization costs | Through study completion, an average of 1 year
  Patients in the virtual stoma group who did not have a second surgery due to complications recorded the costs after low anterior resection for rectal cancer, if the virtual stoma group required bedside or secondary surgery for diverting ileostomy due to complications and all patients in the diverting ileostomy group required reoperation for stoma reversal, record the costs due to complications and reoperation since the data of low anterior resection for rectal cancer.

OTHER OUTCOMES:
Whether patients undergo terminal ostomy after low anterior resection for rectal cancer. | Through study completion, an average of 1 year
  Hartmann's procedure or for example, abdominoperineal extirpation
Patients with stoma (terminal/loop) at 6 months after initial surgery | 6 months from the date of low anterior resection for rectal cancer
  Patients carrying stoma 6 months after low anterior resection for rectal cancer.
The number of participants with virtual ileostomy converted to diverting ileostomy | Through study completion, an average of 1 year
  The virtual stoma required bedside or secondary surgery for diverting ileostomy due to complications.
The number of patients who required secondary abdominal surgery under general anesthesia due to complications | Through study completion, an average of 1 year
  Patient undergoes second abdominal surgery for complications after first surgery
Ghost ileostomy remove time | During hospitalization,approximately 7 days
  Duration of days from the date of radical resection of rectal cancer to virtual stoma removed.
The number of patients with complications after low anterior resection for rectal cancer | Through study completion, an average of 1 year
  Abdominal abscess,Anastomotic bleeding,Pelvic infection,Surgical incision infection, Peritonitis,Interventional drainage ,ileostomy wounds/abscesses/edema/dermatitis/ ulcers,Parastomal hernia ,Stoma prolapse,Anastomotic separation/poor healing, Anastomotic stenosis,Anastomotic leakage,Bowel obstruction,Anastomotic bowel necrosis ,Wound dehiscence / bleeding / sinus tract / abscess/fat liquefaction,Acute kidney injury ,Dehydration/output >1500 mL/day,Converted to permanent ileostomy,Intestinal fistula,Incisional hernia ,fecal incontinence.
Adjuvant chemotherapy in patients after low anterior resection for rectal cancer. | 6 months from the date of low anterior resection for rectal cancer
  Whether the patient has completed chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: fan li, Principal Investigator — Daping Hospital, Third Military Medical University
Locations (2):
- China (2):
  - Daping hospital, Chongqing
  - Daping Hospital, Third Military Medical University, Chongqing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Degiuli M, Elmore U, De Luca R, De Nardi P, Tomatis M, Biondi A, Persiani R, Solaini L, Rizzo G, Soriero D, Cianflocca D, Milone M, Turri G, Rega D, Delrio P, Pedrazzani C, De Palma GD, Borghi F, Scabini S, Coco C, Cavaliere D, Simone M, Rosati R, Reddavid R; collaborators from the Italian Society of Surgical Oncology Colorectal Cancer Network Collaborative Group. Risk factors for anastomotic leakage after anterior resection for rectal cancer (RALAR study): A nationwide retrospective study of the Italian Society of Surgical Oncology Colorectal Cancer Network Collaborative Group. Colorectal Dis. 2022 Mar;24(3):264-276. doi: 10.1111/codi.15997. Epub 2021 Dec 6. PMID 34816571
- [Background] Zhao S, Zhang L, Gao F, Wu M, Zheng J, Bai L, Li F, Liu B, Pan Z, Liu J, Du K, Zhou X, Li C, Zhang A, Pu Z, Li Y, Feng B, Tong W. Transanal Drainage Tube Use for Preventing Anastomotic Leakage After Laparoscopic Low Anterior Resection in Patients With Rectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2021 Dec 1;156(12):1151-1158. doi: 10.1001/jamasurg.2021.4568. PMID 34613330
- [Background] Chapman WC Jr, Subramanian M, Jayarajan S, Makhdoom B, Mutch MG, Hunt S, Silviera ML, Glasgow SC, Olsen MA, Wise PE. First, Do No Harm: Rethinking Routine Diversion in Sphincter-Preserving Rectal Cancer Resection. J Am Coll Surg. 2019 Apr;228(4):547-556.e8. doi: 10.1016/j.jamcollsurg.2018.12.012. Epub 2019 Jan 9. PMID 30639302
- [Background] Kim JH, Kim S, Jung SH. Fecal diverting device for the substitution of defunctioning stoma: preliminary clinical study. Surg Endosc. 2019 Jan;33(1):333-340. doi: 10.1007/s00464-018-6389-4. Epub 2018 Aug 14. PMID 30109482
- [Background] Tsujinaka S, Suzuki H, Miura T, Sato Y, Shibata C. Obstructive and secretory complications of diverting ileostomy. World J Gastroenterol. 2022 Dec 21;28(47):6732-6742. doi: 10.3748/wjg.v28.i47.6732. PMID 36620340
- [Background] Murken DR, Bleier JIS. Ostomy-Related Complications. Clin Colon Rectal Surg. 2019 May;32(3):176-182. doi: 10.1055/s-0038-1676995. Epub 2019 Apr 2. PMID 31061647
- [Background] Huttner FJ, Probst P, Mihaljevic A, Contin P, Dorr-Harim C, Ulrich A, Schneider M, Buchler MW, Diener MK, Knebel P. Ghost ileostomy versus conventional loop ileostomy in patients undergoing low anterior resection for rectal cancer (DRKS00013997): protocol for a randomised controlled trial. BMJ Open. 2020 Oct 15;10(10):e038930. doi: 10.1136/bmjopen-2020-038930. PMID 33060088
- [Background] Miccini M, Amore Bonapasta S, Gregori M, Barillari P, Tocchi A. Ghost ileostomy: real and potential advantages. Am J Surg. 2010 Oct;200(4):e55-7. doi: 10.1016/j.amjsurg.2009.12.017. PMID 20887836
- [Background] Sacchi M, Legge PD, Picozzi P, Papa F, Giovanni CL, Greco L. Virtual ileostomy following TME and primary sphincter-saving reconstruction for rectal cancer. Hepatogastroenterology. 2007 Sep;54(78):1676-8. PMID 18019692
- [Background] Zenger S, Gurbuz B, Can U, Balik E, Yalti T, Bugra D. Comparative study between ghost ileostomy and defunctioning ileostomy in terms of morbidity and cost-effectiveness in low anterior resection for rectal cancer. Langenbecks Arch Surg. 2021 Mar;406(2):339-347. doi: 10.1007/s00423-021-02089-w. Epub 2021 Feb 4. PMID 33537875
- [Background] Baloyiannis I, Perivoliotis K, Diamantis A, Tzovaras G. Virtual ileostomy in elective colorectal surgery: a systematic review of the literature. Tech Coloproctol. 2020 Jan;24(1):23-31. doi: 10.1007/s10151-019-02127-2. Epub 2019 Dec 9. PMID 31820192